CLINICAL TRIAL: NCT06915441
Title: Lipid Infusions to Optimize Nutrition (LION) and Minimize Bronchopulmonary Dysplasia and Neurodevelopmental Impairment in Extremely Preterm Infants: A Randomized Controlled Trial
Brief Title: Lipid Infusions to Optimize Nutrition Trial
Acronym: LION
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Lindsay Fleig Holzapfel, MD, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HSC-MS-24-1129
Record Dates: First submitted 2025-03-27; First posted 2025-04-08 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Bronchopulmonary Dysplasia; Neurodevelopmental Impairment
Keywords: soybean oil-based lipid emulsion (SOLE); mixed oil lipid emulsion (MOLE)
MeSH Terms: conditions — Bronchopulmonary Dysplasia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- SOLE (Experimental)
  Interventions: Drug: SOLE
- MOLE (Active Comparator)
  Interventions: Drug: MOLE

INTERVENTIONS:
Drug: SOLE — Participants will first receive LE at 1 g/kg/day, then will advance to 2 g/kg/day and lastly to 3 g/kg/day as tolerated to titrate based on triglyceride level <250 mg/dL, per clinical team
  Arms: SOLE
Drug: MOLE — Participants will first receive LE at 1 g/kg/day, then will advance to 2 g/kg/day and lastly to 3 g/kg/day as tolerated to titrate based on triglyceride level <250 mg/dL, per clinical team
  Arms: MOLE

SUMMARY:
The purpose of this study is to identify survival free of bronchopulmonary dysplasia (BPD), fatty acid profiles, and early biochemical measures for oxidative stress comparing mixed oil lipid emulsion (MOLE) vs soybean oil-based lipid emulsion (SOLE) and to establish whether MOLE or SOLE is more effective in minimizing pulmonary outcomes, neonatal morbidities, long-term morbidity and mortality, and improving discharge growth and Bayley Scales of Infant Development Fourth Edition (BSID-IV) neurodevelopmental assessment at two years

ELIGIBILITY:
Inclusion Criteria:

* inborn <28 weeks gestational age (GA) or ≤1000g birth weight (BW)
* survives until 12 hours after birth.

Exclusion Criteria:

* Infants who are unable to be enrolled by 96 hours postnatal age
* Major anomaly
* Overt non-bacterial infection
* Infants likely to expire soon defined as limiting or withdrawal of intensive care recommended or requested by the parents.

Ages: 12 Hours to 28 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 230 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-07-30 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants free of BPD (infants breathing in room air) | 36 weeks post menstrual age (PMA)

SECONDARY OUTCOMES:
Change in relative mole percentages of Docosahexaenoic acid (DHA) in plasma | baseline before LE exposure, end of the intervention period (28±3 postnatal days), 36 weeks postmenstrual age (±3 days)
Relative mole percentages of Docosahexaenoic acid (DHA) in plasma | baseline before LE exposure
Relative mole percentages of Docosahexaenoic acid (DHA) in plasma | end of the intervention period (28±3 postnatal days)
Relative mole percentages of Docosahexaenoic acid (DHA) in plasma | 36 weeks postmenstrual age (±3 days)
Change in relative mole percentages of Eicosapentaenoic acid (EPA) in plasma | baseline before LE exposure, end of the intervention period (28±3 postnatal days), 36 weeks postmenstrual age (±3 days)
Relative mole percentages of Eicosapentaenoic acid (EPA) in plasma | baseline before LE exposure
Relative mole percentages of Eicosapentaenoic acid (EPA) in plasma | end of the intervention period (28±3 postnatal days)
Relative mole percentages of Eicosapentaenoic acid (EPA) in plasma | 36 weeks postmenstrual age (±3 days)
Change in relative mole percentages of Arachidonic acid (ARA) in plasma | baseline before LE exposure, end of the intervention period (28±3 postnatal days), 36 weeks postmenstrual age (±3 days)
Relative mole percentages of Arachidonic acid (ARA) in plasma | baseline before LE exposure
Relative mole percentages of Arachidonic acid (ARA) in plasma | end of the intervention period (28±3 postnatal days)
Relative mole percentages of Arachidonic acid (ARA) in plasma | 36 weeks postmenstrual age (±3 days)
Change in relative mole percentages of linoleic acid (LA) in plasma | baseline before LE exposure, end of the intervention period (28±3 postnatal days), 36 weeks postmenstrual age (±3 days)
Relative mole percentages of linoleic acid (LA) in plasma | baseline before LE exposure
Change in relative mole percentages of linoleic acid (LA) in plasma | end of the intervention period (28±3 postnatal days)
Change in relative mole percentages of linoleic acid (LA) in plasma | 36 weeks postmenstrual age (±3 days)
Change in Urine oxidative stress marker, superoxide dismutase | baseline before LE exposure, end of the intervention period (28±3 postnatal days), 36 weeks postmenstrual age (±3 days)
Change in Urine oxidative stress marker, lipid peroxidase | baseline before LE exposure, end of the intervention period (28±3 postnatal days), 36 weeks postmenstrual age (±3 days)
Change in glutathione ratio | baseline before LE exposure, end of the intervention period (28±3 postnatal days), 36 weeks postmenstrual age (±3 days)
Amount of superoxide dismutase | baseline before LE exposure
Amount of superoxide dismutase | end of the intervention period (28±3 postnatal days)
Amount of superoxide dismutase | 36 weeks postmenstrual age (±3 days)
Glutathione ratio | baseline before LE exposure
Glutathione ratio | end of the intervention period (28±3 postnatal days)
Glutathione ratio | 36 weeks postmenstrual age (±3 days)
Amount of lipid peroxidase | baseline before LE exposure
Amount of lipid peroxidase | end of the intervention period (28±3 postnatal days)
Amount of lipid peroxidase | 36 weeks postmenstrual age (±3 days)
Change in lung reactance as assessed by the Non-Invasive Functional Oscillometry Test (FOT) | before discharge (~ 36 weeks post menstrual age), two years
Change in resistance as assessed by the Non-Invasive Functional Oscillometry Test (FOT) | before discharge (~ 36 weeks post menstrual age), two years
Change in impedance as assessed by the Non-Invasive Functional Oscillometry Test (FOT) | before discharge (~ 36 weeks post menstrual age), two years
Change in resonance frequency as assessed by the Non-Invasive Functional Oscillometry Test (FOT) | before discharge (~ 36 weeks post menstrual age), two years
Change in tidal volume as assessed by the Non-Invasive Functional Oscillometry Test (FOT) | before discharge (~ 36 weeks post menstrual age), two years
Change in respiratory rate as assessed by the Non-Invasive Functional Oscillometry Test (FOT) | before discharge (~ 36 weeks post menstrual age), two years
Change in weight of participant | baseline, end of the intervention period (28±3 postnatal days), 36 weeks postmenstrual age, at discharge (~ 40 weeks post menstrual age)
Change in length of participant | baseline, end of the intervention period (28±3 postnatal days), 36 weeks postmenstrual age, at discharge (~ 40 weeks post menstrual age)
Change in head circumference of participant | baseline, end of the intervention period (28±3 postnatal days), 36 weeks postmenstrual age, at discharge (~ 40 weeks post menstrual age)
Neurodevelopmental development as assessed by the Bayley Scales of Infants Development Version IV (BSID-IV) | 2 years corrected age
  The following domains will be assessed: composite motor, language and cognition.Range of composite score is from 40-160.Composite scores (mean = 100; Standard Deviation = 15) will be reported, with higher scores reflecting better developmental outcomes.
Mechanical ventilation days | Discharge (about 3 months from birth)
Number of days participants are exposed to oxygen | Discharge (about 3 months from birth)
Number of chronic lung disease re-hospitalizations | after Neonatal Intensive Care Unit (NICU) discharge till 2 years of age
Number of participants that develop late onset sepsis | Discharge (about 3 months from birth)
Number of participants that develop cholestasis | Discharge (about 3 months from birth)
Weight of participant | Discharge (about 3 months from birth)
Length of participant | Discharge (about 3 months from birth)
Head circumference of participant | Discharge (about 3 months from birth)
Number of participants that die | Discharge (about 3 months from birth)
Number of participants that die | at 2 years
Number of participants that develop Neonatal Morbidity | Discharge (about 3 months from birth)
  Neonatal Morbidity may include severe intraventricular hemorrhage, surgical necrotizing enterocolitis (stage 2A or greater), severe retinopathy of prematurity (Stage 2 or greater or with plus disease), hearing loss, severe bronchopulmonary dysplasia or death.

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Holzapfel, MD, MS, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No